CLINICAL TRIAL: NCT06105554
Title: Phase I/II Open Label Study of Belumosudil Mesylate Alone, and in Combination With Dexamethasone, in Patients With Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi US Services, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0527; NCI-2023-09082 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (dose escalation) (Experimental): Phase 1, the dose of belumosudil mesylate participants receive will depend on when participants join this study. The first group of participants will receive the lowest dose level of belumosudil mesylate.
  Interventions: Drug: Belumosudil mesylate
- Phase 2 (dose expansion) (Experimental): Phase 2, participants will receive belumosudil mesylate at the recommended dose that was found in Phase 1.
  Interventions: Drug: Belumosudil mesylate

INTERVENTIONS:
Drug: Belumosudil mesylate — Given by PO

SUMMARY:
Phase 1 is to find the recommended dose of belumosudil mesylate that can be given to patients with relapsed/refractory MM.

Phase 2 is to learn if the dose of belumosudil mesylate found in Phase 1 can help to control the disease.

DETAILED DESCRIPTION:
Primary Objectives:

* In Phase I, define the toxicities and recommended Phase II dose (RP2D) of belumosudil mesylate in a population of patients with relapsed/refractory multiple myeloma.
* In Phase II, obtain preliminary evidence of efficacy of belumosudil mesylate and further expand the safety experience in this patient population. The overall response rate (ORR) will be defined using the International Myeloma Working Group Uniform Response Criteria as the proportion of patients who, on an intent-to-treat basis, achieve at least a partial response (PR) or better on either belumosudil mesylate alone, or with dexamethasone.
* In Phase II, obtain preliminary evidence of efficacy of the combination of belumosudil mesylate with dexamethasone, with the ORR defined as above.

Secondary Objectives:

* Examine the clinical benefit response rate (CBR), defined as patients experiencing at least a minimal response (MR) or better on belumosudil mesylate alone, and on belumosudil mesylate with dexamethasone.
* Examine the disease stabilization rate (DSR), defined as patients experiencing at least stable disease (SD) or better on belumosudil mesylate alone, and on belumosudil mesylate with dexamethasone.
* Determine durability of responses to single agent belumosudil mesylate, and/or in combination with dexamethasone, including the progression free survival (PFS), minimal residual disease (MRD) negativity in patients achieving a very good partial remission (VGPR) or complete response (CR), duration of response (DOR), and time to next treatment (TTNT).
* Compare the MRD, response, and durability of therapy in patients with standard- and high-risk disease defined by FISH.
* Evaluate the impact of therapy and symptom burden with single agent belumosudil mesylate alone, and of belumosudil mesylate with dexamethasone, on patients with relapsed/refractory multiple myeloma on patient-reported outcomes using the European Organization for Research on the Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core 30 (QLQ-C30).

Exploratory/Correlative Study Objectives:

* The baseline bone marrow sample will be separated into CD138+ and CD138- fractions, and the former will be examined by single cell RNA sequencing (scRNA-Seq) and singe cell B-cell receptor sequencing (scBCR-Seq). Also, the CD138- fraction will be examined by scRNA-Seq, scBCR-Seq, and singe cell T-cell receptor sequencing (scTCR-Seq). Our exploratory objectives are to characterize the myeloma cell's transcriptomic profile, including expression levels of ROCK1 and ROCK2, as well as activation status of the IL-6 pathway to then correlate these to any responses that will be seen.
* The pre-Cycle 3 bone marrow sample will be similarly processed and analyzed. Our exploratory objectives here will be to characterize the transcriptional changes induced by belumosudil mesylate in the myeloma cells themselves, and also the change in the tumor microenvironment (TME), including in the infiltration by, and activation status of immune effector cells.
* Correlate Th17 and regulatory T-cell activation and interleukin level (IL-4, IL6-, IL-17, IL-21, IL-22, and IL-23) changes in myeloma.
* To explore the utility of a CMMC assay in monitoring myeloma disease burden and response kinetics.
* To explore the potential of MicroOrganoSphereTM (MOS) technology to predict clinical

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had a histologically or cytologically confirmed diagnosis of symptomatic multiple myeloma at the time of their initial diagnosis, which requires the presence of all three of the following criteria:

  * Clonal bone marrow plasma cells ≥10%, AND
  * A monoclonal protein in either the serum or urine (except in subjects with non-secretory myeloma), AND
  * Evidence of end-organ damage or a myeloma-defining event that can be attributed to the underlying plasma cell proliferative disorder (to include one or more of the following):
  * Hypercalcemia (corrected calcium >2.75 mmol/L or 11.5 mg/dL); OR
  * Renal insufficiency attributable to myeloma (serum creatinine > 1.9 mg/dL); OR
  * Anemia; normochromic, normocytic with a hemoglobin value ≥2 g/dL below the lower limit of normal, or a hemoglobin or <10 g/dL; OR
  * Bone lytic lesions, severe osteopenia or pathologic fractures detected on a radiographic boney survey, OR
  * More than 1 myeloma-related lesion on advanced imaging, including either by magnetic resonance imaging (MRI), whole-body MRI (WB-MRI), positron emission tomography with embedded computed tomography (PET/CT), or whole-body low dose computed tomography (WB-LDCT); OR
  * Clonal bone marrow plasma cells ≥60%; OR
  * Involved/uninvolved serum free light chain ratio of 100 or more
* Patients with a biopsy-proven plasmacytoma and either a serum or urine monoclonal protein will also be considered to have met the diagnostic criteria for multiple myeloma in the absence of clonal marrow plasmacytosis of ≥10% but must still meet the criteria for evidence of end-organ damage.
* Patients must have measurable disease, as defined by at least one of the following:

  * Serum monoclonal protein level ≥0.5 g/dL for IgG, IgA, or IgM disease
  * Monoclonal protein or total serum IgD or IgE above the upper limit of normal for IgD or IgE disease
  * Urinary M-protein excretion of ≥200 mg over a 24-hour period if the serum monoclonal protein does not meet the above criteria
  * Involved free light chain level ≥10 mg/dL, along with an abnormal free light chain ratio, if the serum monoclonal protein and urinary monoclonal protein do not meet the above criteria
  * Bone marrow involvement of at least 30% if none of the above criteria are met
* Patients must have measurable refractory/relapsed multiple myeloma for which they have received three (3) or more prior lines of therapy with triple class (proteasome inhibitor (PI), immunomodulatory drug (IMiD), and anti-CD38 monoclonal antibody (mAb)) refractory disease. This study will also allow patients who may be double class refractory and intolerant to a third class that precludes administration of that agent, such as neuropathy precluding PI use, allergies to IMiDs, or infusion/injection reactions to CD38 mAbs. Radiation therapy, corticosteroids, or both must have been completed at least 2 weeks prior to the administration of the first dose of belumosudil mesylate. Concurrent use of corticosteroids for conditions other than myeloma are allowed, providing that the total daily dose does not exceed 7.5 mg of prednisone, or its equivalent if a different corticosteroid is being used.
* Patients must be age 18 or older, must be willing and able to provide voluntary written informed consent, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2 (Appendix 13.5), unless the performance status is 3 due to disease burden or disease-related symptoms, such as pain.
* Patients must have evidence of adequate bone marrow reserves, as defined by the following:

  * Absolute neutrophil count (ANC) ≥1,000 cells/mm3 without growth factor support within 1 week of the initiation of treatment
  * Total white blood cell count (WBC) ≥2,000 cells/mm3 without growth factor support within 1 week of the initiation of treatment
  * Hemoglobin ≥8 g/dL without red blood cell transfusions within 2 weeks of the initiation of treatment
  * Platelet count of ≥50,000 cells/mm3
* Patients must have evidence of adequate hepatic function, as defined by the following:

  * Total bilirubin ≤2.5 times the institutional upper limit of the normal values (IULN), except for patients that have previously suspected Gilbert's disease
  * Total aspartate aminotransferase (AST (SGOT)) and alanine aminotransferase (ALT (SGPT)) ≤2.5 times the IULN
* Patients must have evidence of adequate cardiac function, as defined by the following:

  * Absence of New York Heart Association (NYHA) class II, III, or IV congestive heart failure (Appendix 13.6)
  * Absence of uncontrolled angina or hypertension
  * Absence of myocardial infarction in the previous 6 months
  * Absence of clinically significant bradycardia, or other uncontrolled cardiac arrhythmia, defined as grade 3 or 4 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
  * Corrected QT interval (QTc) <480 milliseconds using Fridericia's QT correction formula (QTc = QT / RR1/3)
* Patients must have evidence of adequate renal function, as defined by the following:

  * Serum creatinine within the institutional normal limits, OR if the creatinine is elevated
  * Creatinine clearance (CrCl) ≥30 mL/min., as measured by a 24-hour urine collection, or estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (CKD-EPI) equation (43) as follows:
  * eGFRcr = 142 x min(Scr/κ, 1)α x max(Scr/κ, 1)-1.200 x 0.9938Age x 1.012 [if female], where:
  * Scr = standardized serum creatinine in mg/dL
  * κ = 0.7 (females) or 0.9 (males)
  * α = -0.241 (female) or -0.302 (male)
  * min(Scr/κ, 1) is the minimum of Scr/κ or 1.0
  * max(Scr/κ, 1) is the maximum of Scr/κ or 1.0
  * Age (years)
* HIV seropositive patients with acceptable organ function who meet the patient selection criteria, and who are not on combination anti-retroviral therapy, and who have an absolute CD4+ count >1,000 cells/mm3 of blood, will be eligible.
* Male patients must agree to use an adequate method of contraception for the duration of the study since the effects of belumosudil mesylate on the developing human fetus are unknown. Female patients must be either post-menopausal, free from menses for ≥2 years, surgically sterilized, or willing to use two adequate barrier methods of contraception to prevent pregnancy or must agree to abstain from heterosexual activity throughout the study. Female patients of childbearing potential must have a negative serum (HCG) or urine pregnancy test before receiving the first dose of belumosudil mesylate. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients who are receiving any concurrent investigational agent with known or suspected activity against multiple myeloma, or those whose adverse events due to chemotherapeutic/ immunologic agents or radiation therapy administered more than 2 weeks earlier have not recovered to a severity of grade 0 or grade 1, or to their pre-treatment baseline.
* Patients who have an ECOG >2 will be excluded from this clinical trial because of their poor functional status which could confound the evaluation of adverse events unless this is felt to be disease-related and not from comorbid medical conditions.
* Patients with a known history of allergic reactions attributed to compounds of similar chemical or biologic composition to belumosudil mesylate.
* Patients with known clinically active hepatitis A, B, and/or C infection, due to the difficulty that would be faced in assessing the attribution of any events of hepatic toxicity while on belumosudil mesylate therapy. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Uncontrolled intercurrent illness including not related to multiple myeloma, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, in the opinion of the Principal Investigator.
* The effects of belumosudil mesylate on the developing human fetus are unknown, and women of child-bearing potential and men must therefore agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (follicle stimulating hormone and estradiol in menopausal range, or women who have received whole pelvic radiation therapy).
  * History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device (IUD), tubal ligation or hysterectomy, subject/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant, or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of belumosudil mesylate administration.
* Pregnant or lactating women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with belumosudil mesylate. Male patients with female partners who could potentially become pregnant, will not be excluded but will be required to pursue contraceptive methods.
* Patients with a "currently active" second malignancy should not be enrolled. Patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for >5 years, and are considered by their physician to be at less than 30% risk of relapse. Finally, patients who are on hormonal therapy for a history of either prostate cancer or breast cancer may enroll, provided that there has been no evidence of disease progression during the previous three years.
* Patients with active plasma cell leukemia, defined as having ≥5% of peripheral white blood cells comprised of CD138+ plasma cells (44), or known POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
* Patients who have required plasmapheresis and exchange less than 2 weeks prior to initiation of therapy with belumosudil.
* Patients who are HIV positive and on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with belumosudil mesylate. However, HIV seropositive patients with acceptable organ function who meet the patient selection criteria, and who are not on combination antiretroviral therapy, will be eligible.
* Patients who have known and currently active central nervous system involvement with multiple myeloma will be excluded from this clinical trial because of their poor prognosis, and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Orlowski, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org